CLINICAL TRIAL: NCT02142348
Title: Longitudinal Study of Primary Osteoporosis in Shanghai Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Cui xuejun, Vice director, Shanghai University of Traditional Chinese Medicine
Other Study IDs: Shanghai OP Survey
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Primary Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Basal whole blood is collected for serum and DNA extraction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- osteoprosis research

SUMMARY:
To popularize knowledge of prevention and health care of osteoporosis.To investigate the prevalence of primary osteoporosis in community residents.

DETAILED DESCRIPTION:
1. Objective:

   * To popularize knowledge of prevention and health care of osteoporosis.
   * To investigate the prevalence of primary osteoporosis in community residents.
2. Method:

   * The survey study included the five boroughs of six communities in Shanghai (Xuhui District 2, Pudong New Area 1, Minhang District 1, Pudong New Area 1, Jiading District 1). 10,000 participants are expected to be included.
   * Through a questionnaire and physical examination form, carries on the investigation to the 50-85 years old postmenopausal women during the 3-year follow-up period.
   * Make a survey of Bone Mineral Density,SF-36,international osteoporosis foundation ONE-MINUTE OSTEOPOROSIS RISK TEST,Markers of bone metabolism test,EQ-5D,Hepatic-renal function test and thyroid stimulating hormone level test.
   * Physicians in each community as the backbone, Shanghai University of Traditional Chinese Medicine, Longhua Hospital is responsible for personnel training.
   * Shanghai Clinical Research Center is responsible for program and data management.
   * Shanghai District Health and Family Planning Commission is responsible for coordinating the organization.

ELIGIBILITY:
Inclusion Criteria:

* Had clinical diagnosis of osteoporosis.
* With Bone Mineral Density by dual energy X-ray examination, T value <-2.5 or less.
* Be willing to and be able to join in the study and signed Informed consent.

Exclusion Criteria:

* Excluding the impact of endocrine diseases of bone metabolism (gonadal, adrenal, parathyroid and thyroid disease), rheumatoid arthritis and other autoimmune diseases that affect the absorption of calcium and vitamin D and regulation of the digestive tract and kidney disease, multiple myeloma and other malignant diseases, long-term use of corticosteroids or other drugs affecting bone metabolism, and a variety of congenital and acquired diseases of bone metabolism.
* if they were unable to complete the study survey.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomly selected two communities in Xuhui District to investigate.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density | baseline

SECONDARY OUTCOMES:
SF-36 | baseline
  a composite of functional status
international osteoporosis foundation ONE-MINUTE OSTEOPOROSIS RISK TEST | baseline
Markers of bone metabolism test | baseline
  Fasting peripheral blood collected 2ml.Markers of bone metabolism test，including alkaline phosphatase, 25-hydroxy-vitamin D，prepeptide typeⅠ procollagen，osteocalcin，type I collagen cross-linked C-terminal telopeptide，tartrate resistant acid phosphatase.
EQ-5D | baseline
  A standardised instrument for use as a measure of health outcome.
Hepatic-renal function test | baseline
  Fasting peripheral blood collected 2ml.Hepatic-renal function test，including calcium, phosphorus, creatinine.
thyroid stimulating hormone level test | baseline
  Fasting peripheral blood collected 1ml for thyroid stimulating hormone test.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Dr, Principal Investigator — Study Principal Investigator Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu H, Zhang H, Aimaiti R, Yuan C, Cai F, Wang H, Ji J, Liang J, Cui J, Wang J, Shu B, Xu H, Liang Q, Shi Q, Sun Q, Fang R, Tang D, Wang Y; China Community-based Cohort of Osteoporosis (CCCO) collaborative group. Early-life malnutrition exposure associated with higher osteoporosis risk in adulthood: a large-scale cross-sectional study. Int J Surg. 2025 Jan 1;111(1):190-199. doi: 10.1097/JS9.0000000000002057. PMID 39196877